CLINICAL TRIAL: NCT05161208
Title: Randomized, Controlled, Double-masked Investigator Initiated Study to Evaluate the Efficacy of OC-01 (Varenicline) Nasal Spray on Objective and Subjective Dry Eye Signs and Symptoms in Daily Disposable Contact Lens Wearers
Brief Title: OC-01 (Varenicline) Nasal Spray and Dry Eye Signs and Symptoms in Daily Disposable Contact Lens Wearers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center for Ophthalmic and Vision Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP-001
Record Dates: First submitted 2021-11-30; First posted 2021-12-17 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- OC-01 (varenicline 0.6mg/ml) nasal spray (Experimental): Intranasal delivery of OC-01 nasal spray twice daily (BID)
  Interventions: Drug: OC-01 (varenicline 0.6mg/ml) Nasal Spray
- Placebo (vehicle) nasal spray (Placebo Comparator): Intranasal delivery of placebo vehicle nasal spray twice daily (BID)
  Interventions: Drug: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: OC-01 (varenicline 0.6mg/ml) Nasal Spray — Intranasal delivery of OC-01 nasal spray twice daily (BID)
  Arms: OC-01 (varenicline 0.6mg/ml) nasal spray
Drug: Placebo (vehicle) nasal spray — Intranasal delivery of Placebo (vehicle) nasal spray twice daily (BID)
  Arms: Placebo (vehicle) nasal spray

SUMMARY:
This study is a single center, prospective, randomized, controlled, double-masked, two-arm investigator-initiated study to investigate the efficacy of OC-01 (varenicline) nasal spray on the signs and symptoms of dry eye disease in daily soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed written consent prior to study-related procedures.
2. Be ages 18 to 70 3. Is a symptomatic CL wearer with a CLDEQ-8 score of ≥12 points at baseline at the end of wear time.

4. Soft contact lens wearers with self-reported complaints of dryness and/or reduced contact lens wear time.

5. Wear soft contact lenses 2 or more days a week for more than 1 month in both eyes.

6. Currently wears daily soft lenses in both eyes, for a minimum of 2 days/week for 6 hours/day over the last month, and is willing to continue to do so during the study.

7. Have a current contact lens prescription. 8. Best corrected visual acuity of 20/25-2 or better in each eye (Can achieve acceptable lens fit as well as visual acuity (VA) correctable to logMAR +0.10 or better in each eye with their habitual contact lens type).

9. History or current use of artificial tears at least once in the last 30 days.

10. Be literate and able to complete questionnaires independently. 11. Be able and willing to use the study drug and participate in all study assessments and visits.

12. Have sufficient hand strength, in the opinion of the Investigator, to be able to independently administer the study drug.

13. Have provided written informed consent. 14. If a female is of childbearing potential, they must not plan to get pregnant during the study.

Exclusion Criteria:

1. Wearing soft CLs on an extended wear basis (i.e. overnight) or is a rigid gas permeable lens or hybrid lens wearer
2. Patients with dry eye complaints that the investigator deems are not related to dry eyes will be discontinued at Visit 1.
3. Using prescription eyedrops for the treatment of dry eye disease (ex. Steroids, Lifitegrast, Cyclosporine)
4. Clinically significant ocular trauma.
5. Active or Inactive ocular Herpes simplex or Herpes Zoster infection
6. Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) at the discretion of the investigator.
7. Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye).
8. Severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
9. Eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis).
10. Ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, map dot fingerprint dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity).
11. Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
12. Have had nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
13. Be currently treated with nasal continuous positive airway pressure
14. Have any untreated nasal infection at Visit 1
15. Have a vascularized polyp, severely deviated septum, chronic recurrent nosebleeds, or severe nasal obstruction.
16. Have current concomitant use of a nicotinic acetylcholine receptor agonist [Nicoderm®, Nicorette®, Nicotrol NS® (nicotine), Tabex®, Desmoxan® (cytisine), and Chantix® (varenicline)] within the previous 30 days of Visit 1 and during the treatment period.
17. Use of topical presecription ophthalmic medications including cyclosporine, liftegrast, steroids, non-steroidal anti-inflammatory drugs, anti-glaucoma medications within 7 days of screening or during study period.
18. Prescription and OTC ophthalmic mast cell stabilizers and antihistamines within 21 days of screening and throughout study period (systemic permitted.)
19. Have a known hypersensitivity to any of the procedural agents or study drug components
20. Have active or uncontrolled, severe at the discretion of the investigator: (a) Systemic allergy, (b) Chronic seasonal allergies at risk of being active during the study treatment period, (c) Rhinitis or sinusitis requiring treatment such as antihistamines, decongestants, oral or aerosol steroids at the Screening Visit or be expected to require treatment during the treatment period of the study
21. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1 and during the treatment period.
22. Be a female who is pregnant, nursing, or planning a pregnancy at Visit 1. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
CLDEQ-8 scores at 4 weeks | 4 weeks
  Mean change in CLDEQ-8 scores from baseline to week 4
Contact lens wear time at 4 weeks | 4 weeks
  Mean change in comfortable wear time, overall wear time, and utilization of artificial tears from baseline to week 4 as measured by virtual daily log

SECONDARY OUTCOMES:
CLDEQ-8 scores at 8 weeks | 8 weeks
  Mean change in CLDEQ-8 scores from baseline overtime through Week 8
Contact lens wear time at 8 weeks | 8 weeks
  Mean change in comfortable wear time, overall wear time, and utilization of artificial tears from baseline overtime through Week 8 as measured by virtual daily log
Automated tear breakup time | 8 weeks
  Mean change of automated tear film surface quality breakup time (TFSQ-BUT) over contact lenses from baseline overtime through week 8
Tearscope tear breakup time | 8 weeks
  Mean change in non-invasive tear break up time (NIBUT) from baseline overtime through week 8 as measure and rated by Tearscope Plus
Vital staining score | 8 weeks
  Mean change in vital staining overall score after lens removal from baseline overtime to week 8 as measured by masked evaluator

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Ophthalmic and Vision Recearch, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No